CLINICAL TRIAL: NCT00230607
Title: A Multicenter, Multinational Study of the Effects of Fabrazyme (Agalsidase Beta) Treatment on Lactation and Infants
Brief Title: Study of the Effects of Fabrazyme Treatment on Lactation and Infants
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Per FDA decision, the 2003 Post Marketing commitment has been fulfilled.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGAL02603; 2006-001910-33 (EudraCT Number); MSC12868 (Other: Sanofi)
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Fabry Disease; Alpha Galactosidase A Deficiency
Keywords: alpha Galactosidase A; aGAL; r-haGAL; Fabry; GL3; Fabrazyme; Lysosomal Storage Disorder; Enzyme Replacement Therapy (ERT)
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases | interventions — agalsidase beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fabrazyme (Experimental): Mothers with Fabry disease who received commercially available Fabrazyme intravenous infusion as part of the standard of care while lactating/pregnant and their infants who were breastfed while the mothers were receiving Fabrazyme were enrolled in this study.
  Interventions: Drug: agalsidase beta

INTERVENTIONS:
Drug: agalsidase beta — Pharmaceutical form: powder for reconstitution Route of administration: intravenous
  Other Names: r-haGAL; Fabrazyme

SUMMARY:
The study was planned for up to 2 years (24 months). Planned full participation for both mother and infant was 24 months, planned full participation of mother and development of infant was 24 months, while planned full participation of mother and no infant participation was 6 months.

ELIGIBILITY:
Inclusion Criteria:

Mothers that met the following criteria were enrolled in this study:

* provided signed written informed consent to participate in this study,
* be enrolled in the Fabry Registry and received Fabrazyme while lactating,
* agreed to adhere to the Fabry Registry recommended schedule of assessments for medical history, pregnancy outcome, genotyping, and antibody testing, and
* agreed to adhere to the schedule of evaluations for this study.

Infants that met the following criteria were enrolled in this study:

* had the signed written informed consent of the parent(s)/legal guardian(s) to participate in this study,
* born to a mother who was receiving Fabrazyme during lactation,
* received breast milk from the mother, and
* had the agreement of the parent(s)/legal guardian(s) to adhere to the schedule of evaluations for this study.

Exclusion Criteria:

* The mother and infant were excluded from this study if the mother received an investigational drug within 30 days prior to study enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-05-28 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Investigational Site Number 840005, Decatur, Georgia
  - Investigational Site Number 840006, Fairfax, Virginia
  - investigational site number 01Rhead, Milwaukee, Wisconsin
- investigational site number 04Bodamer, Marl, Austria
- investigational site number 03Waldek, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 active sites in 3 countries. A total of 7 participants were enrolled from 28 May 2006 to 04 March 2022 in this study.
Pre-assignment Details: Mothers/pregnant women enrolled in Fabry Registry, who had received Fabrazyme during lactation/pregnancy and infants born to mother who were receiving Fabrazyme during lactation period were enrolled in this study. This is a rare disease study, with very few participants enrolled. Based on the low enrollment number, the study was terminated by the Sponsor. Overall Arm has been reported in participant flow, Baseline and AE section to protect and maintain participant privacy/confidentiality.
Groups:
- Fabrazyme: Mothers with Fabry disease who received commercially available Fabrazyme intravenous infusion as part of the standard of care while lactating/pregnant, and their infants who were breastfed while the mothers were receiving Fabrazyme were enrolled in this study.
Period: Overall Study
Arm/Group | Fabrazyme
Started | 7
Completed | 4
Not Completed | 3
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Fabrazyme
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Alpha-galactosidase (αGAL) in Plasma
Description: Plasma concentration of αGAL was analyzed. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Month 1, 3, and 6
Population: Evaluable data was collected for 3 participants only; and thus, was not presented to protect participant confidentiality.
Groups:
- Mothers: Mothers with Fabry disease who received commercially available Fabrazyme intravenous infusion at the prescribed dose and regimen as part of the standard of care while lactating/pregnant as determined by their treating physician were enrolled in this study.
Arm/Group | Mothers
Number analyzed (Participants) | 0

2. Primary Outcome: Concentration of Alpha-galactosidase in Breast Milk
Description: Concentration of αGAL in breast milk was analyzed. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Month 1, 3, and 6
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

3. Primary Outcome: Pharmacokinetics: Observed Maximum Plasma Concentration (Cmax) of Alpha-galactosidase A
Description: Cmax was defined as the maximum observed concentration in plasma. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Month 1, 3, and 6
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

4. Primary Outcome: Pharmacokinetics: Observed Maximum Plasma Concentration of Alpha-galactosidase A in Breast Milk
Description: Cmax was defined as the maximum observed concentration in breast milk. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Month 1, 3 and 6
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

5. Primary Outcome: Pharmacokinetics: Area Under the Plasma Alpha-galactosidase A Concentration Versus Time Curve From Time Zero to Two Hours Post End of Infusion (AUC0-2plasma) of Fabrazyme
Description: AUC0-2plasma was defined as the area under the plasma concentration versus time curve from time zero to 2 hours post end of infusion, calculated using the trapezoidal method. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Month 1, 3 and 6
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

6. Primary Outcome: Pharmacokinetics: Area Under the Milk Alpha-galactosidase A Concentration Versus Time Curve From Time Zero to Two Hours Post End of Infusion (AUC0-2milk) of Fabrazyme
Description: AUC0-2milk was defined as the area under the milk concentration versus time curve from time zero to 2 hours post-end of infusion, calculated using the trapezoidal method. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Month 1, 3 and 6
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

7. Primary Outcome: Pharmacokinetics: Lactation Clearance of Alpha-galactosidase A
Description: Lactation clearance was determined in the 0 to 2 hours interval, according to the following equation: the amount of αGAL excreted over the sampling period divided by the AUC during the sampling period. AUC was defined as area under the plasma αGAL concentration-time curve from time 0 to 2 hours post-end of infusion. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Month 1, 3 and 6
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

8. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to 2 Hours (AUC0-2): Milk to Plasma Ratio
Description: AUC0-2milk was defined as the area under the milk concentration versus time curve from time zero to 2 hours post end of infusion, calculated using the trapezoidal method. AUC0-2plasma was defined as the area under the plasma concentration versus time curve from time zero to 2 hours post end of infusion, calculated using the trapezoidal method. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Month 1, 3 and 6
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

9. Primary Outcome: Total Volume of Breast Milk
Description: Collected breast milk samples were analyzed for total volume. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline, Month 2, 6, and 12
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

10. Primary Outcome: Total Fat Content in Breast Milk
Description: Collected breast milk samples were analyzed for total fat content. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline, Month 2, 6, and 12
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

11. Primary Outcome: Total Protein Content in Breast Milk
Description: Collected breast milk samples were analyzed for total protein content. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline, Months 2, 6, and 12
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

12. Primary Outcome: Lactation Status of Mothers at Baseline, Months 1, 2, 3, 4, and 6
Description: Lactation status of mothers was assessed by asking them the question 'Was the infant breastfed?'. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline, Months 1, 2, 3, 4, and 6
Population: as for outcome 1
Arm/Group | Mothers
Number analyzed (Participants) | 0

13. Primary Outcome: Medical History of Enrolled Mothers
Description: Medical history of enrolled mothers collected from Fabry registry. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline
Population: Based on the low enrollment number (5 participants), no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Mothers
Number analyzed (Participants) | 0

14. Primary Outcome: Genotype of the Enrolled Mothers
Description: Genotype of each enrolled mother was collected from the Fabry registry. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline
Population: as for outcome 13
Arm/Group | Mothers
Number analyzed (Participants) | 0

15. Primary Outcome: Pregnancy Outcome
Description: Pregnancy outcome of each enrolled mother collected from the Fabry registry. Baseline for mothers was defined as within 1 month prior to delivery. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline
Population: as for outcome 13
Arm/Group | Mothers
Number analyzed (Participants) | 0

16. Primary Outcome: Number of Mothers Who Were Seropositive for Anti-Fabrazyme Immunoglobulin G (IgG) Antibodies at Baseline
Description: IgG antibodies data of the enrolled mothers were collected from the Fabry registry. Formation or continued presence of serum IgG antibodies to r-haGAL was considered seropositive. Baseline for mothers was defined as within 1 month prior to delivery. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline
Population: as for outcome 13
Arm/Group | Mothers
Number analyzed (Participants) | 0

17. Primary Outcome: Medical History of Infants at Baseline
Description: Medical history of infants included birth difficulties (i.e., normal or caesarian birth). Baseline for infants was at birth. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline
Population: Based on the low enrollment number (2 participants), no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Infants: Infants born to the enrolled mother with Fabry disease who received Fabrazyme during lactation.
Arm/Group | Infants
Number analyzed (Participants) | 0

18. Primary Outcome: Number of Infant Participants With Abnormal Physical Examination
Description: Physical examination of the infants included: length, weight, head circumference, vital signs, general appearance, skin, head, ears, eyes, nose, throat, lymph nodes, heart, lungs, abdomen, extremities/joints, neurological mental status and external genitalia. Baseline for infants was at birth. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline, Months 1, 2, 4, 6, 12, 18 and 24
Population: as for outcome 17
Arm/Group | Infants
Number analyzed (Participants) | 0

19. Primary Outcome: Appearance, Pulse, Grimace, Activity, and Respiration (APGAR) Score of Infants at 1 Minute and 5 Minutes After Birth
Description: The Apgar score is a method to quickly summarize the health of newborn children. The Apgar score is determined by evaluating the newborn baby on five simple criteria: appearance (skin color), pulse (heart rate), grimace (reflex irritability), activity (muscle tone) and respiration on a scale from 0 to 2. Apgar total score (obtained by summing up values from all five items) ranges from 0 to 10 with a score of 0 expressing the worst neonatal status and a score of 10 the best status. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: At 1 minute and 5 minutes after birth
Population: as for outcome 17
Arm/Group | Infants
Number analyzed (Participants) | 0

20. Primary Outcome: Growth Response of Infants
Description: Effects of Fabrazyme on the growth response of infants born to mothers with Fabry disease, who had received fabrazyme during lactation. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Months 1, 2, 3, 6, 12, 18 and 24
Population: as for outcome 17
Arm/Group | Infants
Number analyzed (Participants) | 0

21. Primary Outcome: Development Response of Infants
Description: Effects of Fabrazyme on the development response of infants born to mothers with Fabry disease, who had received fabrazyme during lactation. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Months 1, 2, 3, 6, 12, 18 and 24
Population: as for outcome 17
Arm/Group | Infants
Number analyzed (Participants) | 0

22. Primary Outcome: Number of Infants Seropositive for Anti-Fabrazyme Immunoglobulin G Antibodies
Description: Formation or continued presence of serum IgG antibodies to r-haGAL was considered as seropositive. Baseline for infants was at birth. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline, Months 2, 6, and 12
Population: as for outcome 17
Arm/Group | Infants
Number analyzed (Participants) | 0

23. Primary Outcome: Number of Infants Seropositive for Anti-Fabrazyme Immunoglobulin M Antibodies
Description: Formation or continued presence of serum IgM antibodies to r-haGAL was considered as seropositive. Blood samples of umbilical cord collected immediately after birth was used for the Baseline assessment. Baseline for infants was at birth. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline, Months 2, 6, and 12
Population: as for outcome 17
Arm/Group | Infants
Number analyzed (Participants) | 0

24. Primary Outcome: Genotype of the Infants
Description: Genotype testing was conducted on umbilical cord blood to determine diagnosis of Fabry disease. Baseline for infants was at birth. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline
Population: as for outcome 17
Arm/Group | Infants
Number analyzed (Participants) | 0

25. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAEs)
Description: Adverse event (AE): any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. Serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: From Baseline (Mother: within 1 month prior to delivery; Infant: at birth) up to Month 24
Population: Based on the low enrollment number (7 participants), no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Fabrazyme: Mothers with Fabry disease who received commercially available Fabrazyme intravenous infusion at the prescribed dose and regimen as part of the standard of care while lactating/pregnant as determined by their treating physician were enrolled in this study. Infants born to the enrolled mothers with Fabry disease who received Fabrazyme during lactation were also enrolled.
Arm/Group | Fabrazyme
Number analyzed (Participants) | 0

26. Primary Outcome: Number of Participants Who Received Concomitant Medications
Description: Concomitant medication was any medication, prescription or over-the-counter, taken by a participant during their participation in an investigational study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: From Baseline (Mother: within 1 month prior to delivery; Infant: at birth) up to Month 24
Population: as for outcome 25
Arm/Group | Fabrazyme
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From Baseline (Mother: within 1 month prior to delivery; Infant: at birth) up to Month 24
Description: Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Fabrazyme
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This is a rare disease study, with very few participants enrolled. The study was terminated by the Sponsor. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT00230607/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT00230607/SAP_001.pdf